CLINICAL TRIAL: NCT03497559
Title: Pilot Randomized Controlled Trial on Music Use for Sedation In Critically Ill Children
Brief Title: Music Use for Sedation In Critically Ill Children
Acronym: MUSiCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Women and Children's Health Research Institute, Canada (Other); World Federation of Pediatric Intensive and Critical Care Societies (Unknown)
Responsible Party: Principal Investigator, Gonzalo Garcia Guerra, Associate Profesor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RES0036130
Record Dates: First submitted 2018-03-26; First posted 2018-04-13 (Actual); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Music Therapy; Critical Care; Analgesia; Ventilators, Mechanical
MeSH Terms: conditions — Agnosia | interventions — Music Therapy

STUDY DESIGN:
Intervention Model Description: Double blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: iPods with music and no music, same headphones. Patients and parents are blinded to the intervention the same as bedside nurses, data collectors and principal investigators.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Music (Experimental): Patients will received 30 minutes of classical music 3 times per day . Music will be delivered with noise cancellation headphones.
  Interventions: Other: Music
- Noise cancellation (Sham Comparator): Patients will received 30 minutes of silent recording 3 times per day . Music will be delivered with noise cancellation headphones.
  Interventions: Other: Music
- Control (No Intervention): Patients will receive standard of care.

INTERVENTIONS:
Other: Music — Classical music
  Other Names: Noise cancellation
  Arms: Music; Noise cancellation

SUMMARY:
Stress induced by pain and anxiety is common in pediatric intensive care unit (PICU) patients and can impede the delivery of care as well as their recovery. Sedation/analgesia in PICU is usually achieved using narcotics and benzodiazepines. Excessive use of these drugs can put patients at risk for hemodynamic and respiratory instability, prolonged mechanical ventilation, withdrawal symptoms, and delirium. Non-pharmacologic measures for analgesia and anxiolysis may reduce the total medication requirement and their side effects. The use of non-pharmacologic interventions, including music, has been recommended by sedation guidelines for critically ill patients; however, it is not clear how these interventions should be provided. We plan to conduct a pilot 3-arm RCT to determine the feasibility of a music intervention and assess its effects on sedation/analgesia requirements in children admitted to PICU. Children will be randomly assigned to receive music, noise cancellation or control. Music will be delivered by headphones and an iPod. Music will consist on classical music selected by the study's pediatric music therapist. The noise cancellation group will receive the same headphones but without music. Clinical care of the participants, including use of sedation and analgesia drugs, will not be protocolized. Primary outcomes of this pilot trial is feasibility. Secondary outcomes are drug requirements for sedation and analgesia, and incidence of delirium. These requirements will be captured as a daily intensity score and intermittent dose (PRN) frequency. Mixed-effects models will be used to analyze the effect of the music on sedation/analgesia requirements.

DETAILED DESCRIPTION:
Aim and Objectives Overall Research Question Does music reduce sedation requirements in critically ill children? Purpose statement We plan to conduct a pilot randomized controlled trial (RCT) to determine the feasibility of a pediatric music medicine trial, and to study the effects of music on sedation requirements in children admitted to the pediatric intensive care unit (PICU).

Objectives: a) To demonstrate the feasibility of a music RCT in pediatric critical care; b) To estimate the effect of music on the sedation requirements of critically ill children; c) to obtain information about standard deviation and mean treatment effect for future sample size calculation for a larger trial.

Hypothesis:

We hypothesize that: a) A RCT of music in critically ill children will be feasible; b) Music will result in a 20 % reduction in sedation requirements.

Methodology Study design: We propose a pilot 3 arm RCT. Randomization will be done by a computer-based program to ensure allocation concealment. A total of 30 patients will be randomly assigned in a 1:1:1 ratio to receive music, noise cancellation or control.

Setting: Pediatric Intensive Care Units (Cardiac and General) at the Stollery Children's Hospital, Edmonton, Alberta.

Study Population: critically ill children on mechanical ventilation and receiving sedation and/or analgesia.

Intervention After consent and randomization, patients will be started on the assigned intervention (music/noise cancellation/control) 24-48 hours after admission to the PICU. Based on the neonatal and adult studies, in the music and noise cancellation groups the intervention will be delivered during 30 minutes, at least 3 times a day. The control group will receive usual care. Music will be delivered with the use of noise cancellation headphones and an iPod touch (Apple, California). Music selection will be chosen based on the patient's age. Classical music has been selected by a pediatric music therapist based on its observed properties to settle and calm children. In the noise cancellation group the intervention will be provided with the same headphones connected to an iPod with a silent recording. Children will be assessed with the Sedation behavior scale (SBS) before and during the intervention.29 Signs of agitation or an increase in the SBS will indicate failure of the intervention. Patients will remain on protocol for a maximum of 7 days as long as they are on invasive mechanical ventilation. A parent survey will be conducted at the end of the study. This survey will be conducted on paper or electronically (REDCap, Research Electronic Data Capture) as per the parents' preference.

Concomitant interventions: Clinical care will not be protocolized, and will be according to usual care. Sedative administration will not be directed by the study protocol; it will be up to the attending PICU physician. Assessment of the patients' sedation status and withdrawal symptoms will be conducted every 6 hours by the bedside nurse. Sedation status will be assessed with the use of the SBS while withdrawal will be assessed with the Withdrawal Assessment Tool (WAT-1) score; both are well validated tools .29-32 Demographic variables: To assess if the groups are comparable, including known risk factors, we will record the following: demographic variables (sex, weight, age, diagnosis, operative status, Paediatric Risk of Mortality (PRISM) score, inotrope score, Paediatric logistic organ dysfunction (PELOD) score, baseline SBS, invasive procedures, presence of invasive lines and tubes).

Outcome variables: Feasibility, sedation requirements and delirium. Adverse events Adverse events such as significant negative change in vital signs and/or any other sign of intolerance (agitation) to the intervention will be recorded. We will also record any skin or ear problems (pressure injuries) thought to be associated with the use of headphones.

Study procedures: Patients admitted to the Stollery Children's Hospital PICU and needing mechanical ventilation will be screened for eligibility and approached for consent. After consent, patient demographics will be recorded. Eligible patients will be randomly assigned in a 1:1:1 ratio to the music, the noise cancellation or the control group. During randomization we will stratify patients by age. As a patient qualifies for the trial, a study number and a randomization number will be assigned. Based on the randomization code the research nurse will proceed with one of the interventions, or control, as described above.

Masking: The research nurse will provide the iPods with music or silent recording based on group allocation and will not disclose this information to the healthcare team or the family. However, it is impossible to blind the use of headphones vs. control. The statistician analyzing the data will be blinded to the group allocation.

Sample size justification: The primary outcome used to determine sample size for a future larger RCT is daily Sedation Intensity Score (SIS). The minimal clinically important difference determined by our survey is a reduction in sedation requirements of 20%.8 This pilot study including 10 patients in each group (total 30 patients) will allow us to obtain pediatric information to calculate a sample size for the larger trial.

Analysis Baseline characteristics will be analyzed by descriptive methods. Analysis will be conducted on intention to treat basis and as per protocol. Mixed-effects models will be used to analyze the primary effect of the music on sedation requirements. Statistical tests will be 2-sided with 0.05 level of significance.

Data collection: Variables will be recorded in an anonymized database using REDCap, Research Electronic Data Capture.34

Expected outcomes and Impact This pilot study is a necessary first step toward the conduct of a larger music trial in critically ill children. To obtain funding from major agencies we need to demonstrate the tolerability and feasibility of the intervention and patient recruitment at our centre. This pilot study will also allow formal sample size calculation for a larger trial and will allow us to obtain feedback from major stakeholders including families.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the Stollery Children's Hospital PICU/PCICU.
* Receiving mechanical ventilation for > 24 hours.
* Parental consent

Exclusion Criteria:

* Known hearing deficit
* Major craniotomy-facial abnormality
* Traumatic Brain injury
* Infants < 1 month or < 3 kg.
* Extracorporeal Life Support with neck cannulation.
* Receiving non-invasive mechanical ventilation.
* Nor receiving sedation/analgesia.
* Enrolled in another intervention RCT.

Ages: 1 Month to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of a music intervention study in critically ill children. Feasibility is defined as a consent rate of 70%. | 1 year
  The primary outcomes is feasibility of a music intervention study in critically ill children. In order to determine feasibility we will collect information on: number of eligible patients, number of patients enrolled, rate of enrollment, time to complete participation, protocol adherence and reasons for protocol deviation.
Feasibility of for enrolment music intervention study in critically ill children. | 1 year
  Feasibility of enrolment is defined as an average enrolment of 5 patients per month.
Feasibility of a music intervention study in critically ill children with a protocol adherence of 80%. | 1 year
  Protocol adherence is defined as receiving the allocated intervention for 30 minutes 3 times/day at least 80% of the time patient remains in the study.

SECONDARY OUTCOMES:
Effects of music on sedation requirements measured with the Sedation Intensity Score | 7 days
  Information on sedation. Data on sedation requirements are necessary to calculate the sample size for a future, larger, trial. Sedation requirements will be captured as a daily intensity score and intermittent dose (PRN) frequency. The sedative drug intensity score aggregates the amount of sedation/analgesia from different drug classes using a weight-adjusted dose of each sedative administered during 4-hour time blocks.14 Every sedation amount, for each drug, is placed in quartiles created by using the patient data during the time the patient are involved in the study. The values are then summed over the six 4-hour blocks to obtain the daily score. The Sedation Intensity Score is numeric and has no units.
Effect of music on delirium measured with the Cornell Assessment of Pediatric Delirium (CAPD) instrument | 7 days
  Delirium will be assesed twice a day (as per usual care) with the Cornell Assessment of Pediatric Delirium (CAPD) instrument. Those patients with a score > 9 in two consecutive measurements will be considered to have PICU delirium.34
  critically ill children
Effects of music on sedation requirements measured with Sedation frequency (number of intermittent [PRN] doses) | 7 days
  Dose frequency will be captured by the administration of a (PRN) dose of any of the sedative drugs. This way of capturing sedation requirements enables us to account for the administration of different and non-equivalent types of drugs.14 The unit of measurement is average number of doses/4 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Gonzalo Garcia Guerra, MD, MSc, Principal Investigator — University of Alberta
Locations (1):
- Stollery Children's Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Garcia Guerra G, Joffe A, Sheppard C, Hewson K, Dinu IA, de Caen A, Jou H, Hartling L, Vohra S; Canadian Critical Care Trials Group. Music Use for Sedation in Critically ill Children (MUSiCC trial): study protocol for a pilot randomized controlled trial. Pilot Feasibility Stud. 2020 Feb 25;6:31. doi: 10.1186/s40814-020-0563-x. eCollection 2020. PMID 32128249